CLINICAL TRIAL: NCT04811729
Title: Effectiveness of a Brief Motivational Intervention in Addressing Excessive Alcohol Consumption in Primary Care
Brief Title: Effectiveness of an Intervention in Patients With Excessive Alcohol Consumption
Acronym: ALCO-AP20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Collaborators: Maimonides Institute for Biomedical Research of Cordoba (IMIBIC) (Unknown); Progress and Health Foundation (Unknown); Córdoba and Guadalquivir Health District (Unknown)
Responsible Party: Principal Investigator, Luis A Perula, Doctor in medicine. Collaborating researcher of the project, Hospital Universitario Reina Sofia de Cordoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALCO-AP20
Record Dates: First submitted 2021-03-11; First posted 2021-03-23 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Consumption; Alcohol Use Disorder
Keywords: Alcohol use disorder
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Intervention based on the Motivational Interview, previously receiving a training program
  Interventions: Behavioral: Motivational interview
- Control Group (Active Comparator): Usual care based on a health counci
  Interventions: Behavioral: Medical advice

INTERVENTIONS:
Behavioral: Motivational interview — The participants will apply an approach based on the Motivational Interview (Rollnick, 2008) in patients with excessive alcohol consumption, previously receiving a training program
  Arms: Experimental Group
Behavioral: Medical advice — Usual care
  Arms: Control Group

SUMMARY:
* Main objective: to verify the effectiveness of a brief intervention, based on the motivational interview (MI), in patients with excessive alcohol consumption assisted in Primary Care (PC).
* Design: a multicenter, randomized, cluster-controlled clinical trial with two parallel arms. PC professionals will be randomized to one of the two study groups: 1) Experimental Group (EG): MI-based approach; 2) Control group (CG): usual care. At least 50 family doctors, residents and nurses will participate, recruiting PC patients (n = 394). GE intervention: Training program to acquire specific skills on approaching risky alcohol consumption. It will consist of a workshop, with two video recordings of consultations with simulated standardized patients, before and after it, with each participant receiving formative feedback at the end. -Intervention GC: medical advice that is usually performed in these patients. To measure the knowledge and attitude of professionals in dealing with patients with alcohol consumption, they will fill out a validated questionnaire. In addition, expert evaluators, after viewing the video recordings, will fill out a check-list to check the attitude of each professional, using the EVEM Scale. -Study population: patients ≥14 years of age with risky consumption, detected by the professional in health centers in the province of Córdoba (Spain). Sample size: Assuming a loss rate of 5%, and the "cluster design effect", the number of subjects to be recruited is estimated at 394 (197 / group). Intervention control mechanism: each participant will be audio-recorded with a real patient in a randomly chosen visit, evaluating her skills with the EVEM scale. The follow-up period for each patient will be 12 months, with 4 visits (initial, per month, 3 months, and 6 months) and 4 interleaved telephone contacts. The main outcome variable will be the level of self-reported alcohol consumption and the AUDIT questionnaire score. -Statistical analysis by intention to treat. Descriptive analysis and initial comparability of the groups will be carried out, and the effect of the intervention (dependent variable: abstinence or consumption reduction and AUDIT score) will be evaluated through bivariate and multivariate analysis.

DETAILED DESCRIPTION:
* Design: controlled, cluster-randomized, open-label, two-parallel-arm, multicenter clinical trial. Primary Care professionals will be randomized to one of the two study groups: 1) Experimental Group (EG): they will apply an approach based on Motivational interview (MI), previously receiving a training program. 2) Control group (CG): usual care. They will receive an instructional program in order to avoid the "contamination" effect of the motivational approach. At least 50 professionals (family doctors, residents and nurses) will participate, each of whom will recruit (through opportunistic search) 9-10 PC patients.
* GE intervention: they will receive a 20-hour training program to acquire specific skills on the approach to patients with risky consumption, which will consist of a workshop, with two video recordings of consultations with simulated standardized patients, one before and others after the same, each participant receiving at the end a personalized training feedback.
* CG intervention: they will not receive the training program in MI, instructing them to carry out the medical advice that they usually carry out in these patients (informative model); They will also be videotaped, in order to verify that the approach they carry out is not motivational. On the other hand, both groups will receive an 8-hour workshop on detection, management and approach to the patient with excessive alcohol consumption, based on the recommendations and the action algorithm postulated by the PAPPS. To measure the knowledge and attitude of the professionals of both groups in relation to the approach of the patient with alcohol consumption, they will fill out a questionnaire validated by our group. In addition, expert evaluators, after viewing the video recordings, will fill out a check-list to check the attitude of each professional, using the EVEM Scale, which has been validated by members of our group.
* Material and / or techniques to be used: The information of the participants will be obtained from tools already validated to assess risk alcohol consumption [Alcohol Use Disorder Identification Test (AUDIT), the motivational interview (EVEM questionnaire)] and satisfaction of the doctor-patient (PDRQ-9). In addition, the MCRS scale (Medical Condition Regard Scale) will be used to evaluate the attitude of health workers in the approach to alcohol, which has not been validated in Spanish to date. The Spanish validation process will be carried out by this research group. -Alcohol Use Disorder Identification Test (AUDIT). Tool designed to identify risky alcohol consumption and comprises 10 questions divided into 3 conceptual domains. The first domain assesses recent alcohol consumption and contains 3 questions (frequency of consumption, typical amount and frequency of heavy consumption). The second domain assesses symptoms of dependence through 3 items (loss of control over consumption, increased relevance of consumption and morning consumption) and finally the third domain assesses harmful alcohol consumption through 4 questions (Feeling of guilt after consumption , memory gaps, alcohol-related injuries and environmental concern about consumption). A result equal to or greater than 8 is considered indicative of risky and harmful consumption, as well as a possible dependence on alcohol. -Evaluation Scale of the Motivational Interview (EVEM). 14-item scale with a score of 0 to 4, created and validated by members of our group, to assess encounters between professionals and patients in which MS is used. This scale analyzes: 1) empathy; 2) facilitation for the patient to position himself; 3) works in accordance with the patient; 4) use open questions; 5) perform reflective listening; 6) performs summaries; 7) validate the patient; 8) agreement of change objectives; 9) promotes the design of action / plan with the patient; 10) avoid discord with the patient; 11) develop a maintenance plan with the patient; 12) global spirit: evocation, collaboration, autonomy, understanding.
* Patient-Doctor Relationship Questionnaire (PDRQ-9). 9-question scale that assesses the doctor-patient relationship in clinical practice. Likert-type scale with 5 categories: 1 ("not at all appropriate"), 2 ("somewhat appropriate"), 3 ("appropriate"), 4 ("quite appropriate") and 5 ("very appropriate"). This scale has been validated in Spanish and will allow knowing the satisfaction of the patient in the alcohol approach developed by the health worker. -Medical Condition Regard Scale (MCRS). 11-question scale that assesses the attitude of health workers in the clinical approach. It is a Likert-type scale with 6 categories (1 = totally disagree, 6 = totally agree). It will be validated in Spanish by our research team.
* Location: Health Centers of the Andalus Health Service of the province of Córdoba (Spain).
* Study population: patients aged 14 or over with risky alcohol consumption (28 Standard Drink Units -SDU- / week in men and 17 SDU / week in women) users of PC services.
* Sample size: the main evaluation criterion will be the self-reported consumption by the patient. Based on a previous study carried out by members of our team, and to detect a difference of 20% between the percentage of patients in abstinence (partial or total) between the EG (37%) and the CG (20%); for an alpha error of 5%, a statistical power of 80%, the size would be 220 subjects (110 / group). Assuming a 5% loss rate and being a cluster randomization system, we will take into account the "design effect". Estimates of the intra-cluster correlation coefficient (ICC) in CCT by cluster in PC show that they are generally less than 0.05. This ICC translates, for a cluster size of 15, into a design effect that corresponds to a factor of 1.7. Assuming this value, the size would be 394 subjects to be recruited (197 in each group).
* Randomization: The randomization unit will be the healthcare professional and the intervention unit will be the patient. Professionals will be assigned randomly and equally (1:1) to one of the two study groups. -Mechanism of control of the interventions: each participant will also be videotaped with a real patient in a visit chosen at random, also evaluating her skills with the EVEM scale.
* The follow-up period for each patient will be 6 months, with 4 visits (initial, per month, at 3 months, and at 6 months), in addition to four interleaved telephone contacts. -Study variables: The main outcome variable will be the level of self-reported alcohol consumption (UBEs) and the score of the Alcohol Use Disorder Identification Test (AUDIT) questionnaire.

ELIGIBILITY:
1. -Inclusion criteria: 1.1.-Present risk alcohol consumption (28 Standard Drink Units -SDU- / week in men and 17 SDU / week in women 1.2.-Present 14 years or more; 3) consent to participate in the clinical trial.
2. -Exclusion criteria: 2.1.Present health problems that prevent the intervention or its follow-up.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | 12 months
  Self-reported alcohol consumption level
AUDIT | 12 months
  Alcohol Use Disorder Identification Test (AUDIT) questionnaire score
Alcohol Use Disorder Identification Test (AUDIT) questionnaire score | 12 months
  Tool designed to identify risky alcohol consumption and comprises 10 questions divided into 3 conceptual domains. The first domain assesses recent alcohol consumption and contains 3 questions (frequency of consumption, typical amount and frequency of heavy consumption). The second domain assesses symptoms of dependence through 3 items (loss of control over consumption, increased relevance of consumption and morning consumption) and finally the third domain assesses harmful alcohol consumption through 4 questions (Feeling of guilt after consumption , memory gaps, alcohol-related injuries and environmental concern about consumption). A result equal to or greater than 8 is considered indicative of risky and harmful consumption, as well as a possible dependence on alcohol.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Angel Fernández García, Doctor, Principal Investigator — Andaluz Health Service
Locations (1):
- Distrito sanitario Córdoba y Guadalquivir, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No